CLINICAL TRIAL: NCT06466759
Title: VideolaryngOscopy With Mc Grath™ vs Direct LaryngosCopy for the Positioning of A Double lumeN endOtracheal Tube (VOLCANO Study)
Brief Title: Videolaryngoscopy vs Direct Laryngoscopy for Double Lumen Tube Lumen Tube Placement - A Multicentre Randomized-controlled Trial (VOLCANO Study)
Acronym: VOLCANO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luca Brazzi (Other)
Collaborators: A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other)
Responsible Party: Sponsor-Investigator, Luca Brazzi, Full Professor, Clinical Director, University of Turin, Italy
Organization: University of Turin, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 915.982
Record Dates: First submitted 2024-06-05; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: One Lung Ventilation; Intubation Complication
Keywords: videolaryngoscope; double-lumen tube; one-lung ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOLCANO - double lumen tube placement with direct laryngoscopy (No Intervention): Patients will receive double lumen tube placement with direct laryngoscopy
- VOLCANO - double lumen tube placement with videolaryngoscopy (Active Comparator): Patients will receive double lumen tube placement with videolaryngoscopy
  Interventions: Device: Mc Grath Videolaryngoscope

INTERVENTIONS:
Device: Mc Grath Videolaryngoscope — Use of Videolaryngoscope with Mc Grath versus direct laryngoscopy
  Arms: VOLCANO - double lumen tube placement with videolaryngoscopy

SUMMARY:
The general aim of the study is to observe whether the use of the Mc Grath™ videolaryngoscope instead of direct laryngoscopy can represent, as in the case of the single-lumen tube, an added value in the placement of the double-lumen tube for surgical procedures involving one-lung ventilation, making intubation on the first attempt more likely and quicker. Secondary objectives include evaluating the presence of an advantage of the Mc Grath™ videolaryngoscope over direct laryngoscopy for the correct placement of the double-lumen tube, the need for additional maneuvers during the intubation procedure, and the presence of intra- and post-procedural complications.

DETAILED DESCRIPTION:
Placement of the double-lumen tube (DLT) can be more challenging because the endobronchial tube is larger (thus worsening glottic view) and more rigid (increasing the risk of trauma and reducing maneuverability during placement). An anatomically easy airway can become more demanding when there's a need to place a double-lumen tube. Success rates and intubation times can vary significantly. The superiority of videolaryngoscopy (VLS) over direct laryngoscopy (DL) is clear regarding the placement of the single-lumen endotracheal tube (SLT). Its use is now "recommended" as the first attempt in anticipated difficult airways and "suggested" for all routine intubations. To date, 19 prospective randomized controlled trials have compared the effectiveness of six VLS devices for DLT intubation versus DL in patients with anticipated non-difficult airways. Key endpoints included glottic view, intubation time, success rate, intubation difficulty rating, incidence of malpositioning, postoperative sore throat, hoarseness, procedure-related complications, and intubation-related stress response. Apart from a superior glottic view with VLS compared to DL, consistent results have not emerged across different studies. This heterogeneity may be attributed to differences in the experience of the operators involved, the type of VLS used, and finally the definition of the primary endpoint. Conducting a randomized controlled study with adequate and larger sample size than previous ones and a homogeneous population can ascertain whether VLS can represent, as in the case of SLT, an added value in DLT placement, guiding clinicians towards its routine use.

It is worth noting that current guidelines on DLT intubation do NOT recommend the "1st choice" use of VLS, a recommendation already existing for SLT placement. For this reason, in clinical practice, both devices are effectively used interchangeably, largely based on individual clinician preferences, which moreover possess comparable expertise in both direct laryngoscopy and videolaryngoscopy.

Aim: To compare the effectiveness of a single videolaryngoscope, the Mc Grath™, versus direct laryngoscopy in placing the double-lumen tube in surgery.

Experimental design: Multicentric Randomized Controlled Trial Primary endpoint: evaluation of the advantage of the Mc Grath™ videolaryngoscope over direct laryngoscopy for double-lumen tube intubation.

Secondary endpoints: Evaluation of the advantage of the Mc Grath™ videolaryngoscope over direct laryngoscopy for intra- and post-procedural complications, need for additional maneuvers, and correct placement of the double-lumen tube.

Study duration: 24 months

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* General anesthesia
* One-lung ventilation via double-lumen tube

Exclusion Criteria:

* Patients who refuse to consent to participation in the study.
* Patients scheduled for awake intubation due to pre-operative evaluation findings of predictors of difficult oxygenation that contraindicate intubation under general anesthesia.
* Patients with anatomical anomalies leading to tracheal and/or laryngeal displacement/compression.
* Patients with contraindications to double-lumen tube placement.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-07-02 (Estimated); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of partecipant with first pass intubation success | up to 1 hour
  first pass intubation success of the Mc Grath™ videolaryngoscope over direct laryngoscopy for double-lumen tube intubation.

SECONDARY OUTCOMES:
Intubation-related complications | 24 hours
  Evaluation of the advantage of the Mc Grath™ videolaryngoscope over direct laryngoscopy for intra- and post-procedural complications, need for additional maneuvers, and correct placement of the double-lumen tube.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT06466759/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT06466759/ICF_001.pdf